CLINICAL TRIAL: NCT03606512
Title: A Randomized, Controlled, Observer-blind, Phase 1/2a Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of Ad26.RSV.preF in RSV-seronegative Toddlers 12 to 24 Months of Age
Brief Title: A Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of Adenovirus Serotype 26 Based Respiratory Syncytial Virus Pre-fusion (Ad26.RSV.Pre-F) Vaccine in RSV-Seronegative Toddlers 12 to 24 Months of Age
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108465; 2017-003859-36 (EudraCT Number); VAC18194RSV2002 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2018-06-20; First posted 2018-07-31 (Actual); Results first posted 2022-11-30 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Syncytial Virus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: RSV Seronegative Toddlers (Ad26.RSV.preF) (Experimental): Respiratory syncytial virus (RSV) seronegative toddlers will receive intramuscular (IM) injection of 2.5*10^10 viral particles (vp) of an adenovirus serotype 26- based vaccine encoding for the respiratory syncytial virus pre-fusion F-protein on Days 1, 29, and 57.
  Interventions: Biological: Ad26.RSV.preF
- Group 2: RSV Seronegative Toddlers (Placebo/Nimenrix) (Placebo Comparator): RSV seronegative toddlers will receive IM injection of placebo on Days 1, 29 and 57. Placebo can be replaced with Nimenrix on Day 57 in countries where applicable.
  Interventions: Biological: Placebo; Biological: Nimenrix

INTERVENTIONS:
Biological: Ad26.RSV.preF — Ad26.RSV.preF will be administered as IM injection at a dose of 2.5*10^10 vp.
  Other Names: JNJ-64400141
  Arms: Group 1: RSV Seronegative Toddlers (Ad26.RSV.preF)
Biological: Placebo — Placebo will be administered as IM injection of sterile 0.9 percent (%) saline for injection.
  Arms: Group 2: RSV Seronegative Toddlers (Placebo/Nimenrix)
Biological: Nimenrix — Nimenrix will be administered as 0.5 milliliter (mL) solution for IM injection.
  Arms: Group 2: RSV Seronegative Toddlers (Placebo/Nimenrix)

SUMMARY:
The purpose of this study is to assess the safety and reactogenicity of an intramuscular regimen of 3 doses of 2.5*10^10 viral particles (vp) of adenovirus serotype 26 based respiratory syncytial virus pre-fusion protein (Ad26.RSV.preF) vaccine in RSV-seronegative toddlers aged 12 to 24 months.

DETAILED DESCRIPTION:
RSV is considered the most important cause of serious acute respiratory illness in children under 5 years of age. Ad26.RSV.preF (JNJ-64400141) investigational vaccine is a replication-incompetent serotype 26 adenoviral vector (Ad26) containing a deoxyribonucleic acid (DNA) transgene that encodes for the F protein derived from the respiratory syncytial virus (RSV) A2 strain stabilized in the pre-fusion conformation (Ad26.RSV.preF). The study will evaluate whether Ad26.RSV.preF is safe, well-tolerated, and immunogenic in RSV-seronegative toddlers. The study will have 3 phases: a screening phase (up to 6 weeks before the first dose), a vaccination phase (34 weeks), and a safety follow-up phase through 2 RSV seasons after the first dose. RSV infection will be monitored by active and passive surveillance. The total duration of the study will be approximately 26 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant who is seronegative for respiratory syncytial virus (RSV) within 42 days prior to dosing
* Participant is the product of a normal term pregnancy greater than or equal to (>=)37 weeks, with a minimum birth weight of 2.5 kilogram (kg)
* Participant must be in good health without any significant medical illness on the basis of physical examination, medical history, and vital signs performed at screening
* Participant has received all routine immunizations appropriate for his or her age according to local guidelines
* Each participant's parent(s)/legal guardian(s) must have access to a consistent means of contact either by telephone contact or email/computer

Exclusion Criteria:

* Participant's weight is below tenth percentile according to World Health Organization (WHO) pediatric growth and weight charts
* Participant has any clinically significant acute or chronic medical condition (for example, history of seizure disorders, bleeding/clotting disorder, autoimmune disease, active malignancy, systemic infections, congenital heart disease, history of any pulmonary condition requiring medication, atopy, reactive airway disease, medically-confirmed wheezing, bronchoconstriction or treatment with a beta 2 agonist, cystic fibrosis, bronchopulmonary dysplasia, chronic pulmonary disease, medically-confirmed apnea, hospitalization for respiratory illness, or mechanical ventilation for respiratory illness) that, in the opinion of the investigator, would preclude participation
* Participant is in receipt of, or planning to receive, live attenuated vaccine (for example, measles, mumps and rubella [MMR] or varicella, but excluding rotavirus vaccine) within 28 days of each study vaccination (that is, before and after); other vaccines (for example, influenza, pertussis, polio or rotavirus) should be given at least 14 days before or 14 days after each study vaccination
* Participant has known or suspected immunodeficiency, such as known human immunodeficiency virus (HIV) infection
* Participant has a known allergy to vaccines or vaccine components (including any of the constituents of the study vaccine), or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine components (including any of the constituents of the study vaccine). Participants with egg allergies can be enrolled

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (25):
- Australia (3):
  - Barwon Health, Geelong
  - Telethon Kids Institute, Nedlands
  - Murdoch Children's Research Institute, Parkville
- Brazil (4):
  - Complexo Hospital de Clinicas - UFPR, Curitiba
  - Hospital Pequeno Principe, Curitiba
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da PUCRS, Porto Alegre
- Canada (4):
  - Dalhousie University, Halifax, Nova Scotia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - McGill University Health Centre - Vaccine Study Centre, Pierrefonds, Quebec
  - CHU de Quebec Universite Laval, Québec, Quebec
- Finland (3):
  - Järvenpään rokotetutkimusklinikka, Jarvenpaa
  - Tampereen rokotetutkimusklinikka, Tampere
  - Turun rokotetutkimusklinikka, Turku
- Poland (2):
  - Jerzy Brzostek Prywatny Gabinet Lekarski, Dębica
  - Szpital im Swietej Jadwigi Slaskiej Oddzial Pediatryczny z Pododdzialem Niemowlecym, Trzebnica
- Spain (4):
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
- Sweden (2):
  - Sachsska barn-och ungdomssjukhuset, Stockholm
  - Norrlands Universitetssjukhus, Umeå
- United Kingdom (3):
  - Imperial College London, London
  - Royal Manchester Children's Hospital, Manchester
  - University Hospital Southampton NHS Foundation Trust, Southampton

REFERENCES:
- [Derived] Langley JM, Nolan TM, Ramet M, Richmond PC, Rosario Filho N, Haazen W, van den Berg SPH, Williams K, Bastian AR, Omoruyi E, Williams Durkin J, Salisch N, Van Geet G, van Duijnhoven W, Heijnen E, Callendret B. A Phase 1/2a Study Evaluating Safety and Immunogenicity of Ad26.RSV.preF in RSV-seronegative Toddlers Aged 12-24 Months. Open Forum Infect Dis. 2024 Aug 8;11(9):ofae453. doi: 10.1093/ofid/ofae453. eCollection 2024 Sep. PMID 39220658

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Nimenrix: Respiratory syncytial virus (RSV) seronegative toddler participants aged greater than or equal to (>=) 12 months to less than or equal to (<=) 24 months received placebo (matching to Ad26.RSV.preF) as an intramuscular (IM) injection on Days 1, 29 and 57. For participants in whose countries the commercial vaccine Nimenrix was licensed, placebo was replaced with Nimenrix as IM injection on Day 57 in accordance with local label and local regulations and based on joint parent/legal guardian and principal investigator (PI) decision.
- Ad26.RSV.preF: RSV seronegative toddler participants aged >=12 months to <=24 months received Ad26.RSV.preF (0.25 mL of 2.5*10^10 viral particles [vp]) as an IM injection on Days 1, 29, and 57.
Period: Overall Study
Arm/Group | Placebo/Nimenrix | Ad26.RSV.preF
Started | 18 | 20
Participants Received Placebo on Day 57 | 6 | 0
Participants Received Nimenrix on Day 57 | 12 | 0
Completed | 18 | 18
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — 'moved from study area | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Nimenrix | Ad26.RSV.preF | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Continuous [Median (Full Range); unit: months] | 18.5 [12 to 22] | 15 [12 to 23] | 16.5 [12 to 23]
Age, Customized [Count of Participants; unit: Participants]
  From 12 months to 24 months | 18 | 20 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 16 | 17 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 13 | 16 | 29
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRALIA | 6 | 8 | 14
  BRAZIL | 2 | 3 | 5
  CANADA | 3 | 2 | 5
  FINLAND | 5 | 6 | 11
  POLAND | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic Adverse Events (AEs) for 7 Days After First Vaccination
Description: An AE is any untoward medical event that occurs in a participants administered an investigational product, and it does not necessarily indicate only events with a clear causal relationship with the relevant investigational product. Solicited local and systemic AEs were precisely defined events that participants were specifically asked about and which were noted by participants in the diary. Solicited local AEs included injection-site pain/tenderness, injection-site erythema and injection-site swelling/induration. Solicited systemic AEs included fatigue, headache, nausea, myalgia and fever.
Time Frame: Up to Day 8 (7 days after first vaccination on Day 1)
Population: The Full Analysis set (FAS) included all participants who were randomized and received at least one dose of study vaccine (placebo or nimenrix, and Ad26.RSV.preF), regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Groups:
- Ad26.RSV.preF: RSV seronegative toddler participants aged >=12 months to <=24 months received Ad26.RSV.preF (0.25 milliliters [mL] of 2.5*10^10 viral particles [ vp]) as an IM injection on Days 1, 29, and 57.
Arm/Group | Placebo/Nimenrix | Ad26.RSV.preF
Number analyzed (Participants) | 18 | 20
Participants
  Solicited Local AEs | 2 | 6
  Solicited Systemic AEs | 11 | 17

2. Primary Outcome: Number of Participants With Solicited Local and Systemic AEs for 7 Days After Second Vaccination
Description: as for outcome 1
Time Frame: Up to Day 36 (7 days after second vaccination on Day 29)
Population: The FAS included all participants who were randomized and received at least one dose of study vaccine (placebo or nimenrix, and Ad26.RSV.preF), regardless of the occurrence of protocol deviations.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Nimenrix | Ad26.RSV.preF
Number analyzed (Participants) | 18 | 20
Participants
  Solicited Local AEs | 1 | 9
  Solicited Systemic AEs | 9 | 11

3. Primary Outcome: Number of Participants With Solicited Local and Systemic AEs for 7 Days After Third Vaccination
Description: as for outcome 1
Time Frame: Up to Day 64 (7 days after third vaccination on Day 57)
Population: The FAS included all participants who were randomized and received at least one dose of study vaccine (placebo or nimenrix, and Ad26.RSV.preF), regardless of the occurrence of protocol deviations. Here, 'N' (Number of participants analyzed) included number of participants evaluable for this outcome measure. Data for this outcome measure was planned to be collected and analyzed per the administered study vaccination type.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Respiratory syncytial virus (RSV) seronegative toddler participants aged greater than or equal to (>=) 12 years to less than or equal to (<=) 24 months received placebo (matching to Ad26.RSV.preF) as an intramuscular (IM) injection on Days 1, 29 and 57.
- Nimenrix: Participants received Nimenrix as an IM injection on Day 57 based on joint parent/legal guardian and PI decision, in countries where the commercial vaccine Nimenrix was licensed.
Arm/Group | Placebo | Nimenrix | Ad26.RSV.preF
Number analyzed (Participants) | 6 | 12 | 19
Participants
  Solicited Local AEs | 1 | 4 | 7
  Solicited Systemic AEs | 3 | 4 | 12

4. Primary Outcome: Number of Participants With Unsolicited AEs for 28 Days After First Vaccination
Description: An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with a clear causal relationship with the relevant investigational product. Unsolicited AEs were precisely defined events that participants were not asked about and which were not noted by participants in the diary.
Time Frame: Up to Day 29 (28 days after first vaccination on Day 1)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Nimenrix | Ad26.RSV.preF
Number analyzed (Participants) | 18 | 20
Participants | 5 | 9

5. Primary Outcome: Number of Participants With Unsolicited AEs for 28 Days After Second Vaccination
Description: An AE is any untoward medical event that occurs in a participants administered an investigational product, and it does not necessarily indicate only events with a clear causal relationship with the relevant investigational product. Unsolicited AEs were precisely defined events that participants were not asked about and which were not noted by participants in the diary.
Time Frame: Up to Day 57 (28 days after second vaccination on Day 29)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Nimenrix | Ad26.RSV.preF
Number analyzed (Participants) | 18 | 20
Participants | 7 | 9

6. Primary Outcome: Number of Participants With Unsolicited AEs for 28 Days After Third Vaccination
Description: as for outcome 5
Time Frame: Up to Day 85 (28 days after third vaccination on Day 57)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants received placebo by intramuscular (IM) injection on Days 1, 29 and 57.
- Nimenrix: Participants received Nimenrix as an IM injection on Day 57 in countries where the commercial vaccine Nimenrix was licensed and based on joint parent/legal guardian and PI decision.
Arm/Group | Ad26.RSV.preF | Placebo | Nimenrix
Number analyzed (Participants) | 19 | 6 | 12
Participants | 7 | 3 | 3

7. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of participants with SAEs were reported. An AE is any untoward medical event that occurs in a participants administered an investigational product, and it does not necessarily indicate only events with a clear causal relationship with the relevant investigational product. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a suspected transmission of any infectious agent via a medicinal product, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Up to 2 year 10 months
Population: The FAS included all participants who were randomized and received at least one dose of study vaccine (placebo or nimenrix, and Ad26.RSV.preF), regardless of the occurrence of protocol deviations. Data for this outcome measure was planned to be collected and analyzed per the administered study vaccination type.
Measure: Count of Participants; unit: Participants
Arm/Group | Ad26.RSV.preF | Placebo | Nimenrix
Number analyzed (Participants) | 20 | 6 | 12
Participants | 1 | 0 | 0

8. Secondary Outcome: Titers of Neutralizing Antibodies to Respiratory Syncytial Virus (RSV) A2 Strain
Description: Neutralizing antibody titers assessed by virus neutralizing antibodies (VNA) against the RSV A2 strain were expressed as 50% inhibitory concentration (IC50) units.
Time Frame: Days 1, 8, 85, and 267 (End of first RSV season)
Population: The Per-protocol Immunogenicity (PPI) analysis set included all randomized and vaccinated participants for whom immunogenicity data are available, excluding participants with major protocol deviations expecting to impact the immunogenicity outcomes. Here, 'n' (number analyzed) included number of participants evaluable for specified time points. Here, values below the seropositivity cut-off (less than [<] 42.7) were imputed with zero.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Placebo/Nimenrix | Ad26.RSV.preF
Number analyzed (Participants) | 18 | 19
Titers
  Day 1 | NA [NA to NA] — Here, NA signifies that Geometric mean and 95% CI were not estimable due to being below lower limit of quantification (LLOQ) of 42.7. | NA [NA to NA] — Here, NA signifies that Geometric mean and 95% CI were not estimable due to being below LLOQ of 42.7.
  Day 8: number analyzed (Participants) | 17 | 18
  Day 8 | NA [NA to NA] — Here, NA signifies that Geometric mean and 95% CI were not estimable due to being below LLOQ of 42.7. | NA [NA to 52] — Here, NA signifies that Geometric mean and 95% CI were not estimable due to being below LLOQ of 42.7.
  Day 85: number analyzed (Participants) | 16 | 14
  Day 85 | NA [NA to 45] — Here, NA signifies that Geometric mean and 95% CI were not estimable due to being below LLOQ of 42.7. | 293 [240 to 358]
  Day 267 (End of first RSV season): number analyzed (Participants) | 15 | 9
  Day 267 (End of first RSV season) | NA [NA to 46] — Here, NA signifies that Geometric mean and 95% CI were not estimable due to being below LLOQ of 42.7. | 269 [115 to 632]

9. Secondary Outcome: Pre-Fusion A Immunoglobulin G (IgG) Serum Antibody Response as Assessed by Enzyme-linked Immunosorbent Assay (ELISA)
Description: Pre-fusion A IgG serum antibody response was assessed by ELISA.
Time Frame: Days 1, 8, 85, and 267 (End of first RSV season)
Population: The PPI analysis set included all randomized and vaccinated participants for whom immunogenicity data are available, excluding participants with major protocol deviations expecting to impact the immunogenicity outcomes. Here, 'n' (number analyzed) included number of participants evaluable for specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units per liter (EU/L)
Arm/Group | Placebo/Nimenrix | Ad26.RSV.preF
Number analyzed (Participants) | 18 | 19
ELISA units per liter (EU/L)
  Day 1 | NA [NA to NA] — Here, NA signifies that Geometric mean and 95% CI were not estimable due to being below LLOQ of 16.1. | NA [NA to NA] — Here, NA signifies that Geometric mean and 95% CI were not estimable due to being below LLOQ of 16.1.
  Day 8: number analyzed (Participants) | 17 | 19
  Day 8 | NA [NA to NA] — Here, NA signifies that Geometric mean and 95% CI were not estimable due to being below LLOQ of 16.1. | NA [NA to NA] — Here, NA signifies that Geometric mean and 95% CI were not estimable due to being below LLOQ of 16.1.
  Day 85: number analyzed (Participants) | 16 | 14
  Day 85 | NA [NA to NA] — Here, NA signifies that Geometric mean and 95% CI were not estimable due to being below LLOQ of 16.1. | 236 [187 to 299]
  Day 267 (End of first RSV season): number analyzed (Participants) | 15 | 9
  Day 267 (End of first RSV season) | NA [NA to 27] — Here, NA signifies that Geometric mean and 95% CI were not estimable due to being below LLOQ of 16.1. | 212 [79 to 571]

10. Secondary Outcome: Post-Fusion A IgG Serum Antibody Response as Assessed by ELISA
Description: Post-fusion A IgG serum antibody response as assessed by ELISA was reported.
Time Frame: Days 1, 8, 85, and 267 (End of first RSV season)
Population: The PPI analysis set included all randomized and vaccinated participants for whom immunogenicity data are available, excluding participants with major protocol deviations expecting to impact the immunogenicity outcomes. Here, 'n' (number analyzed) is number of participants evaluable for specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/L
Arm/Group | Placebo/Nimenrix | Ad26.RSV.preF
Number analyzed (Participants) | 18 | 19
EU/L
  Day 1 | NA [NA to NA] — Here, NA signifies that Geometric mean and 95% CI were not estimable due to being below LLOQ of 17.0. | NA [NA to NA] — Here, NA signifies that Geometric mean and 95% CI were not estimable due to being below LLOQ of 17.0.
  Day 8: number analyzed (Participants) | 16 | 19
  Day 8 | NA [NA to NA] — Here, NA signifies that Geometric mean and 95% CI were not estimable due to being below LLOQ of 17.0. | NA [NA to NA] — Here, NA signifies that Geometric mean and 95% CI were not estimable due to being below LLOQ of 17.0.
  Day 85: number analyzed (Participants) | 16 | 14
  Day 85 | NA [NA to NA] — Here, NA signifies that Geometric mean and 95% CI were not estimable due to being below LLOQ of 17.0. | 47 [40 to 54]
  Day 267 (End of first RSV season): number analyzed (Participants) | 15 | 9
  Day 267 (End of first RSV season) | NA [NA to 30] — Here, NA signifies that Geometric mean and 95% CI were not estimable due to being below LLOQ of 17.0. | 58 [22 to 153]

11. Secondary Outcome: T-cell Response (Percent [%]) to RSV F Peptides for T-helper (Th) 1 and Th2 Subtyping as Measured by Flow Cytometry
Description: T-cell response (%) to RSV F peptides for T-helper Th1 and Th2 subtyping as measured by flow cytometry was planned to be assessed. Th1(% of Clusters of differentiation 4 [CD4]+ interferon gamma [IFN-g]+T cells; lower limit(s) of quantification [LLOQ]=0.05%) and Th2 (% of CD4+ interleukin [IL]-4+/IL-13+ and CD40L+T cells; LLOQ=0.07%) responses were determined by intracellular cytokines after RSV F peptide stimulation.
Time Frame: Baseline (Day 1) and Day 85
Population: Data for this outcome measure was not collected due to low number of viable peripheral blood mononuclear cells (PBMC), the positive control in the intracellular cytokine staining (ICS) assay (Staphylococcal enterotoxin B [SEB]) could not be performed.
Arm/Group | Placebo/Nimenrix | Ad26.RSV.preF
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Participants With Severe RSV-lower Respiratory Tract Infection (LRTI)
Description: Number of participants with severe RSV-LRTI were reported.
Time Frame: Up to 2 year 10 months
Population: The Modified Intent-to-treat (mITT) analysis set included participants who were randomized and received at least one dose of study vaccine (placebo or nimenrix, and Ad26.RSV.preF), regardless of the occurrence of protocol deviations and who seronegative at screening but for whom there is an anamnestic response at Day 8.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Nimenrix | Ad26.RSV.preF
Number analyzed (Participants) | 18 | 19
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 year 10 months
Description: The Full Analysis set (FAS) included all participants who were randomized and received at least one dose of study vaccine (placebo or nimenrix, and Ad26.RSV.preF), regardless of the occurrence of protocol deviations. As planned, safety data was summarized per vaccine regimen. Data for adverse events was planned to be collected and analyzed per the administered study vaccination type.
Arm/Group | Placebo | Nimenrix | Ad26.RSV.preF
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/12 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/12 | 1/20
Other Adverse Events (participants affected / at risk) | 6/6 | 8/12 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | Nimenrix (N=12) | Ad26.RSV.preF (N=20)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | Nimenrix (N=12) | Ad26.RSV.preF (N=20)
Middle Ear Effusion (Ear and labyrinth disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Teething (Gastrointestinal disorders) | 0 | 0 | 4
Injection Site Bruising (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Tenderness (General disorders) | 1 | 0 | 0
Allergy to Arthropod Bite (Immune system disorders) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Croup Infectious (Infections and infestations) | 1 | 0 | 2
Exanthema Subitum (Infections and infestations) | 0 | 1 | 0
Hand-Foot-And-Mouth Disease (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 1
Oral Viral Infection (Infections and infestations) | 0 | 0 | 1
Otitis Media (Infections and infestations) | 0 | 3 | 0
Otitis Media Acute (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 5 | 4
Rhinitis (Infections and infestations) | 0 | 0 | 1
Rhinovirus Infection (Infections and infestations) | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 4
Viral Infection (Infections and infestations) | 1 | 0 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 2
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Drooling (Nervous system disorders) | 0 | 0 | 1
Irritability (Psychiatric disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-05-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT03606512/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT03606512/SAP_001.pdf